CLINICAL TRIAL: NCT04936334
Title: The Role of 68Ga-PSMA-11 PET in Surgery Guidance in Prostate Cancer: A Prospective Pilot Trial
Brief Title: The Role of 68Ga-PSMA-11 PET (Prostate Specific Membrane Antigen) in Surgery Guidance in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinton Bahler (Other)
Responsible Party: Sponsor-Investigator, Clinton Bahler, Principal Investigator, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IUSCCC-0760
Record Dates: First submitted 2021-06-11; First posted 2021-06-23 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 68Ga-PSMA-11 PET will be performed and we will study how the knowledge of the results informs treatment decisions versus the treatment decisions with only MRI knowledge.
Masking Description: Two separate radiologists (one from Nuclear Medicine and one from MRI) will read images in a blinded fashion and provide their findings for the surgeons to use in treatment planning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Men diagnosed with clinically significant prostate cancer who are scheduled for prostatectomy (Experimental): 1. Men diagnosed with clinically significant prostate cancer who are scheduled or for prostatectomy will undergo injection of 68Ga-PSMA-11 at the time of their pre-treatment PSMA PET. Followed until 12 mo post surgery
  Interventions: Diagnostic Test: 68Ga-PSMA-11 PET Scan

INTERVENTIONS:
Diagnostic Test: 68Ga-PSMA-11 PET Scan — Patients will undergo injection of 68Ga-PSMA-11 at the time of their pre treatment PSMA PET scan and followed until 12 months post surgery.

SUMMARY:
Obtain PSMA-PET imaging preoperatively and calculate performance for predicting extra-prostatic extension based on whole-mount pathology (gold standard).

Quantify the frequency of proper treatment changes directed by PSMA-PET, focusing on appropriate preservation of surrounding structures important for genito-urinary function including: 1) Bladder neck, 2) Nerve bundles, 3) Urethral Sphincter (Figure 4).

Directly compare PSMA-PET performance for predicting extra-prostatic extension to standard-of-care assessments.

Assess quality of life changes from preoperative baseline.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men diagnosed with clinically significant prostate cancer who are scheduled or scheduling for prostatectomy 2. Prostate pathology results consistent with:

  1. > 3 cores of Gleason 3+4 or
  2. NCCN unfavorable intermediate risk or
  3. NCCN high-risk or
  4. NCCN very-high risk 3. Scheduled for standard of care MRI or has recently completed standard of care MRI (within 6 months).

Willing and able to lie still for approximately 50 minutes in an enclosed space for the PET/CT and MRI

Exclusion Criteria:

* 1. Participation in another investigational trial involving research exposure to ionizing radiation concurrently or within 30 days.

  2. Does not meet safety criteria for MRI scan (e.g. metal implant that could affect prostate imaging).

  3. Significant acute or chronic medical, neurologic, or illness in the subject that, in the judgment of the Principal Investigator, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bahler CD, Tachibana I, Tann M, Collins K, Swensson JK, Green MA, Mathias CJ, Tong Y, Yong C, Boris RS, Brocken E, Hutchins GD, Sims JB, Hill DV, Smith N, Ferari C, Love H, Koch MO. Comparing Magnetic Resonance Imaging and Prostate-Specific Membrane Antigen-Positron Emission Tomography for Prediction of Extraprostatic Extension of Prostate Cancer and Surgical Guidance: A Prospective Nonrandomized Clinical Trial. J Urol. 2024 Aug;212(2):290-298. doi: 10.1097/JU.0000000000004032. Epub 2024 May 24. PMID 38785259

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Prostate lobes (right and left)
Groups:
- PSMA-PET and MRI in Men Scheduled for Prostatectomy: Men diagnosed with clinically significant prostate cancer who are scheduled or for prostatectomy will undergo PSMA PET and MRI.
  There were 100 prostate lobes examined with 2 lobes per patient.
Period: Overall Study
Arm/Group | PSMA-PET and MRI in Men Scheduled for Prostatectomy
Started | 51; 102 Prostate lobes (right and left)
Completed | 50; 100 Prostate lobes (right and left)
Not Completed | 1; 2 Prostate lobes (right and left)
Not completed — Metastatic disease found on PSMA-PET, surgery cancelled | 1

BASELINE CHARACTERISTICS:
Arm/Group | PSMA-PET and MRI in Men Scheduled for Prostatectomy
Number analyzed (Participants) | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.5 [58 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 42
  More than one race | 0
  Unknown or Not Reported | 2
PSA [Median (Inter-Quartile Range); unit: ng/mL] | 7.0 [5.5 to 8.7]
Gleason Grade-group, final pathology [Number; unit: participants] — This is pathology. Prostate cancer uses Gleason grading system, which is organized as the Grade group as follows:
  3+3 = 1, 3+4 = 2, 4+3 = 3, 4+4 = 4, 4+5 = 5,
  Grade group 1 indicates a lower grade cancer.
  participants
    Grade-Group 1 (Gleason) | 1
    Grade-Group 2 (Gleason) | 15
    Grade-Group 3 (Gleason) | 15
    Grade-Group 4 (Gleason) | 9
    Grade-Group 5 | 10
Pathologic stage (T) [Number; unit: participants] — T-stage:
  pT2 (organ confined), pT3a (extra-prostate extension), pT3b (Seminal vesicle invasion), pT4 (outside invasion)
  participants
    pT2 | 25
    pT3a | 12
    pT3b | 13
    pT4 | 0
Pathologic stage (N) [Count of Participants; unit: Participants] — This measure reports the total number of participants with positive lymph nodes. This is also referred to as pathologic N-stage. The N-stage indicates the number of total patients who had positive lymph nodes.
  Participants | 8

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of PSMA-PET and MRI Imaging Preoperatively for Predicting Extra-prostatic Extension
Description: Sensitivity detecting extra-prostatic extension of cancer at the nerve bundles
Time Frame: The patients underwent a 60minute PET exam. The surgery was generally performed within 1month of the PET scan. The pathology was done 5-10 days after the surgery.
Population: Men diagnosed with prostate cancer often seek surgical treatment. Surgical treatment--radical prostatectomy--is currently guided by clinical parameters (PSA, pathology) and MRI imaging. These men often have considerable concerns about the balance of cancer control and quality of life after the surgery. There were 100 prostate lobes examined with 2 lobes per patient. One patient was enrolled but did not complete study procedures.
Measure: Number (95% Confidence Interval); unit: percentage
Units Other Than Participants: prostate lobes
Groups:
- PSMA-PET in Men Diagnosed With Clinically Significant Prostate Cancer Scheduled for Prostatectomy: Men diagnosed with clinically significant prostate cancer who are scheduled or for prostatectomy will undergo injection of 68Ga-PSMA-11 at the time of their pre-treatment PSMA PET. Followed until 12 mo post surgery
  There were 100 prostate lobes examined with 2 lobes per patient.
- MRI in Men Diagnosed With Clinically Significant Prostate Cancer Scheduled for Prostatectomy: Men diagnosed with clinically significant prostate cancer who are scheduled or for prostatectomy will undergo imaging with MRI in addition to PSMA-PET.
  There were 100 prostate lobes examined with 2 lobes per patient.
Arm/Group | PSMA-PET in Men Diagnosed With Clinically Significant Prostate Cancer Scheduled for Prostatectomy | MRI in Men Diagnosed With Clinically Significant Prostate Cancer Scheduled for Prostatectomy
Number analyzed (Participants) | 50 | 50
Number analyzed (prostate lobes) | 100 | 100
percentage | 86 [71 to 100] | 57 [36 to 78]
Statistical Analysis 1: Comparison: PSMA-PET in Men Diagnosed With Clinically Significant Prostate Cancer Scheduled for Prostatectomy vs MRI in Men Diagnosed With Clinically Significant Prostate Cancer Scheduled for Prostatectomy; Test type: Superiority; p < 0.05, McNemar; McNemar = 0.03

2. Primary Outcome: Specificity of PSMA-PET and MRI
Description: Specificity of PSMA-PET and MRI to detect Extra-prostatic extension prior to prostatectomy. Whole mount pathology is used as the reference standard.
Time Frame: Pre-surgery prediction.
Measure: Number (95% Confidence Interval); unit: Percentage
Units Other Than Participants: prostate lobes
Arm/Group | PSMA-PET in Men Diagnosed With Clinically Significant Prostate Cancer Scheduled for Prostatectomy | MRI in Men Diagnosed With Clinically Significant Prostate Cancer Scheduled for Prostatectomy
Number analyzed (Participants) | 50 | 50
Number analyzed (prostate lobes) | 100 | 100
Percentage | 73 [64 to 83] | 77 [68 to 86]

3. Secondary Outcome: 1) Quantify the Frequency of Proper Treatment Changes for Nerve Sparing Directed by PSMA-PET
Description: Rate of treatment changes
Time Frame: 60 Days
Measure: Number; unit: participants
Groups:
- PSMA-PET and MRI in Men Scheduled for Prostatectomy: Men diagnosed with clinically significant prostate cancer who are scheduled or for prostatectomy will undergo PSMA PET and MRI.
Arm/Group | PSMA-PET and MRI in Men Scheduled for Prostatectomy
Number analyzed (Participants) | 50
participants | 20

ADVERSE EVENTS:
Time Frame: 1 day, the day of imaging.
Description: Patient were monitored during injection of the (Ga68)PSMA-11 and afterwards for at least 60minutes.
Arm/Group | PSMA-PET and MRI in Men Scheduled for Prostatectomy
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT04936334/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT04936334/ICF_001.pdf